CLINICAL TRIAL: NCT02123953
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-438 in Healthy Male Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAK-438 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-438/CPH-002; U1111-1153-6907 (Other: World Health Organization)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Dose Finding Study
Keywords: Drug therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- TAK-438 10 mg (Experimental): TAK-438 10 mg, tablets, orally, once, daily, Days 1 to 7.
  Interventions: Drug: TAK-438
- TAK-438 15 mg (Experimental): TAK-438 15 mg, tablets, orally, once, daily, Days 1 to 7.
  Interventions: Drug: TAK-438
- TAK-438 20 mg (Experimental): TAK-438 20 mg, tablets, orally, once, daily, Days 1 to 7.
  Interventions: Drug: TAK-438
- TAK-438 30 mg (Experimental): TAK-438 30 mg, tablets, orally, once, daily, Days 1 to 7.
  Interventions: Drug: TAK-438
- TAK-438 40 mg (Experimental): TAK-438 40 mg, tablets, orally, once, daily, Days 1 to 7.
  Interventions: Drug: TAK-438
- Placebo (Placebo Comparator): TAK-438 placebo-matching tablets, orally, once, daily, Days 1 to 7.
  Interventions: Drug: TAK-438 Placebo

INTERVENTIONS:
Drug: TAK-438 — TAK-438 tablets
  Arms: TAK-438 10 mg; TAK-438 15 mg; TAK-438 20 mg; TAK-438 30 mg; TAK-438 40 mg
Drug: TAK-438 Placebo — TAK-438 placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and pharmacokinetics of TAK-438 following multiple oral doses to healthy adult Japanese male participants

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-438. TAK-438 was being tested to assess side effects and how TAK-438 moves throughout the body after multiple doses have been administered. This study looked at lab results and side effects in people who took TAK-438.

The study consisted of 5 steps covering dose ranges of TAK-438 from 10, 15, 20, 30 and 40 mg once daily for 7 days. The study population for each step included 12 participants. Within each step, 9 participants were randomized to TAK-438 and 3 participants were randomized to placebo. A total of 60 participants were enrolled.

The dosing groups in this study took place in sequential order. Therefore, the TAK-438 15 mg group did not start until the TAK-439 10 mg group had completed, etc. All participants in each dosing group were asked to take the study drug in the morning, after fasting for at least 10 hours, each day throughout the study.

This single-centre trial was conducted in the Japan. The overall time to participate in this study was up to 43 days. Participants made 3 visits to the clinic, including one 11-day period of confinement to the clinic, and a final visit 7 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult Japanese male volunteer.
2. Is 20-45 years old inclusive, at time of giving consent.
3. Is capable of understanding and complying with protocol requirements.
4. Signs a written, informed consent form prior to the initiation of any study procedure.
5. Weighs at least 50 kg and has a body mass index (BMI) of 18.5 to 25.0 kg/m^2 inclusive at screening.
6. Tests negative for hepatitis B surface antigen (HBs), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antigen-antibody and syphilis serum reaction test.
7. The participant who the investigator or subinvestigator confirmed to be eligible to participate in this study based on results of the screening tests, and physical examination, physical findings, vital signs, electrocardiogram (ECG), clinical laboratory tests etc. from 3 days before dosing to before the start of dosing on Day 1 with the study drug.

Exclusion Criteria:

1. Has undergone upper gastrointestinal resectioning or vagetomy.
2. Is judged to have hypoacidity or anacidity.
3. Presently has or a history of acid-related diseases (e.g., erosive esophagitis, duodenal ulcer, gastric ulcer, non-erosive esophagitis, Barrett's esophagitis or Zollinger-Ellison syndrome).
4. Received H. pylori eradication treatment within 6 months prior to the start of treatment with the study drug.
5. Presently has or has a history of hepatic disorder, renal disorder, cardiovascular system disease, blood disease, endocrine disease, metabolic disease, lung disease, gastrointestinal disease, nervous system disease, urological disease, immunological disease or mental illness that makes him not eligible to participate in this study.
6. Presently has or has a history of hypersensitivity or allergy towards drugs or food.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the start of treatment with the study drug.
8. Participant for whom it is difficult to collect blood from the peripheral veins.
9. Has donated more than 200 mL of whole blood within 4 weeks (28 days) or more than 400 mL of whole blood within 12 weeks (84 days) prior to the start of treatment with the study drug.
10. Has donated a total volume of more than 800 mL of whole blood within 52 weeks (364 days) prior to the start of treatment with the study drug.
11. Has given plasma component and plaque component within 2 weeks (14 days) prior to the start of treatment with the study drug.
12. Has used a prescription drug (including over-the counter drugs) within 4 weeks (28 days) prior to the start of treatment with the study drug.
13. Has used vitamins, Chinese herbal remedies, or supplement (including St John's Wort, ginseng, kava kava, ginkgo biloba, melatonin) within 4 weeks (28 days) prior to the start of treatment with the study drug.
14. Has ingested any foods or beverages containing grapefruit (juice or pulp), caffeine, alcohol within 72 hours prior to the start of treatment with the study drug.
15. Administered another study drug within 16 weeks (112 days) prior to the start of treatment with this study drug.
16. Administered TAK-438 in the past.
17. Is considered by the investigator or subinvestigator, for any reason, to be an unsuitable candidate for participating in this study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) | Day 1 to Day 15
  An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it did not necessarily have to have a causal relationship with this treatment. The different categories of intensity (severity) were characterized as follows: Mild: The AE was transient and easily tolerated by the participant.
  Moderate: The AE caused the participant discomfort and interrupted the participant's usual activities. Severe: The AE caused considerable interference with the participant's usual activities.
Number of Participants With Potentially Clinically Significant Vital Sign Findings | Day 1 to Day 15
  Vital signs included blood pressure, pulse, respiratory rate, and body temperature (armpit).
Number of Participants With Potentially Clinically Significant Changes in Body Weight | Day 1 to Day 15
Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings | Day 1 to Day 15
  The investigator or the subinvestigator interpreted the ECG using 1 of the following categories: "within normal limits", "abnormal but not clinically significant", or "abnormal and clinically significant". The time that the ECG was performed was recorded. The following parameters were recorded from the participant's ECG trace: heart rate, RR interval, PR interval, QT interval, QRS duration, and QTc interval.
Number of Participants With Potentially Clinically Significant Laboratory Evaluation Findings | Day 1 to Day 15
  Laboratory tests for hematology, biochemistry, and urinalysis were be performed.
AUC(0-tau): Area Under the Plasma Concentration-time Curve from Time 0 to Time tau Over the Dosing Interval for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  AUC(0-tau) is a measure of the area under the plasma concentration-time curve from the time 0 to time tau over a dosing interval, where tau is the length of the dosing interval, 24 hours, calculated using the linear trapezoidal rule.
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  AUC(0-tlqc) is a measure of the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration, calculated using the linear trapezoidal rule.
AUMC(0-tlqc): Area Under the First Moment Plasma Concentration-time Curve from Time 0 (t1) to Time of the Last Quantifiable Concentration (tlqc) for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  AUMC(0-tlqc) is a measure of the area under the first moment plasma concentration-time curve from time 0 to time of the last quantifiable concentration (tlqc), calculated using the linear trapezoidal rule.
MRT(0-tlqc): Mean Residence Time from Time 0 (t1) to Time of the Last Quantifiable Concentration (tlqc) for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  MRT(0-tlqc) is a measure of the mean residence time from time 0 to time of the last quantifiable concentration (tlqc) calculated as MRT(0-tlqc)=AUMC(0-tlqc)/AUC(0-tlqc).
Cmax: Maximum Observed Plasma Concentration for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  Time to reach the maximum plasma concentration (Tmax), equal to time (hours) to Cmax.
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  AUC(0-inf) is a measure of the area under the plasma concentration-time curve from time 0 to infinity.
Terminal Elimination Rate Constant (λz) for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  Terminal elimination rate constant (λz) is the rate at which drugs are eliminated from the body.
Terminal Elimination Half-life (T1/2) for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  Terminal Phase Elimination Half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Apparent Clearance (CL/F) for TAK-438F | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC(0-24), expressed in L/hr.
Apparent Volume of Distribution (Vz/F) for TAK-438F | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as CL/F divided by λz.
AUMC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  AUMC(0-inf) is a measure of the area under the first moment plasma concentration-time curve from time 0 to infinity.
MRT: Mean Residence Time for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 to 7 predose, Days 1 and 7 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16 hours post- dose, and Day 7 24 hours post-dose
  Mean residence time, calculated as MRT=AUMC(0-inf)/AUC(0-inf)
Cumulative Urinary Excretion Ratio for TAK-438F and TAK-438F metabolites M-I and M-II, M-III and M-IV-Sul | Days 1 predose, and Days 1 and 7 0-6, 6-12, and 12-24 hours post-dose
  The cumulative urinary excretion ratio is defined as the percentage of the dose excreted in the urine.

SECONDARY OUTCOMES:
24-Hour Intragastric pH Profile | Day 1 and Day 7
  To obtain intragastric pH a portable pH measuring device with a miniature glass electrode that was calibrated using standard pH 4 and pH 7 solutions was placed in the stomach transnasally and its positioned confirmed by X-ray guidance. pH data was recorded electronically 8:30 AM to 9:10 AM of the following day every 10 seconds.
Total Amount of Serum Gastrin | Predose Days 1 to 7, Day 7 24 hours post-dose, and Day 15
Total Amount of Serum Pepsinogens I | Predose Days 1 to 7, Day 7 24 hours post-dose, and Day 15
Total Amount of Serum Pepsinogens II | Predose Days 1 to 7, Day 7 24 hours post-dose, and Day 15
Pepsinogens I/Pepsinogens II Ratio | Predose Days 1 to 7, Day 7 24 hours post-dose, and Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

REFERENCES:
- [Derived] Jenkins H, Sakurai Y, Nishimura A, Okamoto H, Hibberd M, Jenkins R, Yoneyama T, Ashida K, Ogama Y, Warrington S. Randomised clinical trial: safety, tolerability, pharmacokinetics and pharmacodynamics of repeated doses of TAK-438 (vonoprazan), a novel potassium-competitive acid blocker, in healthy male subjects. Aliment Pharmacol Ther. 2015 Apr;41(7):636-48. doi: 10.1111/apt.13121. Epub 2015 Feb 23. PMID 25707624